CLINICAL TRIAL: NCT06668935
Title: Prolongation of GLP-1 Adherence When Using Continuous Glucose Monitoring
Status: Recruiting | Type: Observational
Sponsor: Abbott Diabetes Care (Industry)
Responsible Party: Sponsor
Other Study IDs: ADC-US-RES-24254
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Randomization to FSL 3 or Standard of Care: Subjects with type 2 diabetes who are newly beginning GLP-1 or dual GLP-1/GIP drug therapy will be randomized to use either the FSL3 or their existing Standard of Care (SOC) to manage their diabetes.
  Interventions: Device: To utilize the FreeStyle Libre 3 Continuous Glucose Monitoring System (FSL3) to help prolong the length of time people with diabetes maintain adherence to GLP-1 and dual GIP/GLP-1 agonists

INTERVENTIONS:
Device: To utilize the FreeStyle Libre 3 Continuous Glucose Monitoring System (FSL3) to help prolong the length of time people with diabetes maintain adherence to GLP-1 and dual GIP/GLP-1 agonists — All subjects will then begin use of their prescribed GLP-1 or combination GIP/GLP-1 medication in accordance with the HCP's instructions. Subjects will be titrated to their maximum tolerable dose per the medication's approved titration schedule and according to their HCP's standard of care between Visits 2 and 3.

SUMMARY:
This study is to see if the FreeStyle Libre 3 Continuous Glucose Monitoring System (FSL3) will help prolong the length of time people with diabetes maintain adherence to glucagon-like peptide 1 (GLP-1/GIP) agonists.

DETAILED DESCRIPTION:
Subjects with type 2 diabetes who are newly beginning GLP-1 or GLP-1/GIP drug therapy will be randomized to use either FSL3 or their existing Standard of Care to manage their diabetes. Up to 800 subjects will be enrolled across the United States with 200 evaluable subjects in each group (intervention and control) for a total of 400 evaluable subjects. Subjects will be on the study approximately 210 days. Subjects will wear one sensor applied to the back of the upper arm and will have a paired smartphone that will be used to start the sensor and collect glucose readings.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject must be able to read and understand English.
3. Subject must have a type 2 diabetes diagnosis.
4. In the investigator's opinion, subject must meet the criteria for beginning use of GLP-1 or GIP/GLP-1 medications for management of their diabetes.
5. Subject is beginning use of GLP-1 / GIP/GLP-1 medication for management of their diabetes.
6. Subject must be willing to allow venous samples to be obtained to test HbA1c.
7. Subject must be willing to either continue using their existing standard of care device or must be willing to use the FreeStyle Libre 3 Continuous Glucose Monitoring System to manage their diabetes throughout the duration of the study.
8. In the investigator's opinion, the subject must be able to follow the instructions provided to him/her by the study site and perform all study tasks as specified by the protocol.
9. Subject must be available to participate in all study visits.
10. Subject must be willing and able to provide written signed and dated informed consent.

    Exclusion Criteria:
11. Subject is a member of the Study Staff.
12. Subject has a diagnosis of type 1 or gestational diabetes.
13. Subject is currently using or has previously used GLP-1 or GIP/GLP-1 drugs for any reason.
14. Subject is currently using a Continuous Glucose Monitor (CGM) as their standard of care device to manage their diabetes.
15. Subject has known allergy to medical grade adhesive, isopropyl alcohol and/or ethyl alcohol used to disinfect skin.
16. Subject is taking any type of rapid-acting insulin, including Neutral Protamine Hagedorn (NPH) and premix insulin.
17. Subject has concomitant medical condition which, in the opinion of the investigator, could interfere with the study or present a risk to the safety or welfare of the subject or study staff.
18. Subject currently is participating in another clinical trial.
19. Subject is unsuitable for participation due to any other cause as determined by the Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with type 2 diabetes who are newly beginning GLP-1 or dual GLP-1/GIP drug therapy will be randomized to use either the FSL3 or their existing Standard of Care (SOC) to manage their diabetes.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To assess the length of time subjects in each group remain on a GLP-1 or GLP-1/GIP combination drug | 210 days
  The primary outcome is to see if the FreeStyle Libre 3 Continuous Glucose Monitoring System (FSL3) helps prolong the length of time people with diabetes maintain adherence to glucagon-like peptide 1 (GLP-1) and dual gastric inhibitory polypeptide/glucagon-like peptide 1 (GIP/GLP-1) agonists.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Excellence Medical and Research, Miami Gardens, Florida

IPD SHARING:
Plan to Share IPD: Undecided